CLINICAL TRIAL: NCT05316766
Title: Multi-user Touch Surfaces for Promoting Social Participation and Self-efficacy in Upper-limb Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Professor, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMadeira
Record Dates: First submitted 2022-03-02; First posted 2022-04-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Social Interaction; Self Efficacy; Stroke; Motor Activity
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive intervention through the multi-user touch surface
  Interventions: Other: Physical rehabilitation interactive table
- Treatment as usual (Active Comparator): This will receive conventional therapy
  Interventions: Other: Physical rehabilitation

INTERVENTIONS:
Other: Physical rehabilitation — Exercises to rehabilitate upper limb strength, coordination and range of movement, based on conventional therapy
  Arms: Treatment as usual
Other: Physical rehabilitation interactive table — Exercises to rehabilitate upper limb strength, coordination and range of movement, based on multi-user touch surface
  Arms: Intervention

SUMMARY:
The purpose of this study is to compare the efficacy of conventional therapy with a framework intervention for upper limb motor rehabilitation based on the promotion of self-efficacy and social participation/interaction through a multi-user touch surface

DETAILED DESCRIPTION:
After signing the written informed consent about participating in the study, participants will be assessed for exclusion criteria and their motor, social and depression skills prior to intervention. After this, they will undergo a 12 sessions treatment for 4 weeks in groups of three, randomly distributed for a control group and experimental group. At the end of the intervention, participants will be assessed in the same manner as before the intervention. One month after the end of the intervention, participants will be assessed for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivor

Exclusion Criteria:

* Unable to write and read
* Hemispatial neglect
* Previous upper limb motor deficits/lesions that still interfere with function
* History of drugs/alcohol abuse
* Aphasia with difficulties understanding oral communication and/or unability to express orally
* Token equal or under 17
* ARAT score lower than 10 or higher than 54
* Botulinic toxin treatment in the last 4 months
* Beck's Depression Inventory higher than 31

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (change between three time frames ) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Hand Function
Box and Blocks (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Coordination
Dynamometer (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Strength
Nine Hole Peg Test (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Fine motor skills
Motor Activity Log (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Quantity and Quality of movement everyday activities
Reaching Performance Scale in Stroke (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Quality of movement
Fugl-Meyer Assessment (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Range of movement
Stroke Self-Efficacy Questionnaire (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Self-efficacy, minimum 0 maximum 130, higher score means better outcome

SECONDARY OUTCOMES:
Beck's Depression (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Depressive symptoms
Social Interaction category of ''Functional Limitation Profile'' (specific name of the scale) (change between three time frames) | Assessment (before intervention), Reassessment (after 12 x 45 minutes sessions, 3 sessions per week) and Follow-up (1 month after the end of intervention)
  Social Interaction

CONTACTS AND LOCATIONS:
Overall Officials: Sergi B Badia, Principal Investigator — Professor
Locations (1):
- ARDITI, Funchal, Madeira, Portugal

IPD SHARING:
Plan to Share IPD: No